CLINICAL TRIAL: NCT02739204
Title: Development of Novel Diagnostic Tools and Therapeutic Strategies for Oral Cancer
Brief Title: Concurrent Radiotherapy and/or Cisplatin With or Without Celecoxib in Patients With Primary Oral Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Collaborators: Ministry of Health and Welfare, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CMUH102-REC1-071
Record Dates: First submitted 2016-03-22; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Oral Squamous Cell Carcinoma
Keywords: Celecoxib; Relapse-free OSCC patient; Recurrence; Survival; Prognosis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence | interventions — Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Celecoxib (Experimental): Combination of concurrent radiotherapy and/or Cisplatin with or without Celcoxib
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: Celecoxib — 200 mg of Celecoxib daily for 6-month treatment after surgery within 1 - 6 months
  Other Names: Celebrex

SUMMARY:
The research and development of novel anti-tumor agents in oral cancer is slow, the investigation of repositioning use of currently available drugs in clinical, such as a selective cyclooxygenase-2 (COX-2) inhibitor (Celebrex/Celecoxib) maybe a potential alternative strategy.

DETAILED DESCRIPTION:
Celebrex (Celecoxib) is a form of non-steroidal anti-inflammatory drug that directly targets COX-2 enzyme to block the inflammatory signaling and has been approved to treat colon cancer. In our preliminary findings, Celecoxib significantly inhibited cell growth,proliferation, migration, invasion and epithelial-mesenchymal transition programs in oral squamous cell carcinoma cell (OSCC) lines. The Institutional Review Board in China Medical University Hospital (CMUH) has approved the combination treatment of concurrent radiotherapy (RT) and/or Cisplatin with or without Celecoxib in a phase II clinical trial for relapse-free primary OSCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. OSCC patients with T1,2/ N0 and without pathological risk features
2. OSCC patients with T1,2/ N0,1 and pathological risk features
3. OSCC patients with T4a/ N2,3

Exclusion Criteria:

1. Pregnant women paitents
2. Taiwanese aboriginal patients
3. Not primary OSCC patients
4. OSCC patients with dysfunction of liver and/or kidneys

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Relapse-free recurrence | 3 year relapse-free recurrence
  3-year follow-up after 6-month treatment of Celecoxib

SECONDARY OUTCOMES:
Relapse-free survival | 3 year relapse-free survival
  3-year follow-up after 6-month treatment of Celecoxib

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Chin Ko, MD-PhD, Study Chair — Graduate Institute of Clinical Medical Science, China Medical University, Taiwan
Locations (1):
- Department of Otolaryngology, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided